CLINICAL TRIAL: NCT02547181
Title: Comparing Short-term Function and Pain After No Treatment or Splinting for Boxer's Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 341-2014
Record Dates: First submitted 2015-03-06; First posted 2015-09-11 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Metacarpal Fractures
Keywords: Fracture; Follow-up; metacarpal
MeSH Terms: conditions — Fractures, Bone | interventions — Behavior Therapy; Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Splint (Experimental): Patients will be provided instructed to use a tensor bandage as well as specific behaviours to prevent movement of the injured part of the hand.
  Interventions: Behavioral: Splint
- Behavioral Modification (Experimental): Patients are given a removable plaster/fiberglass splint with a tensor bandage underneath
  Interventions: Behavioral: Behavioral Modification

INTERVENTIONS:
Behavioral: Behavioral Modification — Patient will be provided with tensor bandage and instructed on specific behaviors to prevent movement of the injured part of the hand.
  Arms: Behavioral Modification
Behavioral: Splint — fibreglass splint
  Arms: Splint

SUMMARY:
This Study is being done because the investigators would like to know if pain and hand function after having a boxer's fracture differs between being treated with supportive splinting or without splinting, but with behavioral modifications.

DETAILED DESCRIPTION:
After initial treatment in the emergency department, patients with boxer's features are referred to the division of plastic and reconstructive surgery at Sunnybrook hospital. During initial consultation with the hand surgeon, treatment is chosen. Patients are follow-up with their hand surgeon at 4-, 8-, and 12--week intervals.

Supportive splinting: Patient's are given a removable plaster/fiberglass splint with a tensor bandage underneath.

Behavioral Modifications: Patients are not splinted, but provided a tensor bandage. Patients are instructed on specific behaviours to prevent movement of the injured part of the hand.

The purpose of the study is to compare pain and short-term hand function in patients who undergo supportive splinting compared to patients who undergo behavioral modifications treatment only to see which option is associated with shorter functional recovery and which option is associated with less pain during the first 4 weeks after initial treatment.

On follow-up appointments at 4, 8,and 12 weeks, as well as initial consultation with the hand surgeon, participants will be asked to perform a grip strength test with a Jamal Hydraulic hand Dynanometer. Participants will be asked to fill out a Brief Michigan Hand Questionnaire along with the grip strength test as well as quick demographics survey at initial consultation with the hand surgeon. After the 12-week follow up appointment, study participation will end.

If a patient is unable to follow-up with the hand surgeon, the Brief Michigan Hand Questionnaire will be done via phone whenever is most convenient for the patient. It's anticipated that about 40 people will participate in this study at a single centre in Toronto.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of true boxer's fracture
* Candidate for either supportive splinting or tensor bandage
* Speaking, read and write English

Exclusion Criteria:

* Prior surgical treatment for boxer's fractures or other hand conditions.
* Concurrent hand/wrist injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
hand function | 4 weeks
  measured by Brief Michigan Hand Questionnaire (MHQ)
hand function | 8 weeks
  measured by Brief Michigan Hand Questionnaire (MHQ)
hand function | 12 weeks
  measured by Brief Michigan Hand Questionnaire (MHQ)

SECONDARY OUTCOMES:
Grip strength | 4 weeks
  measured using Dynamometer
Grip strength | 8 weeks
  measured using Dynamometer
Grip strength | 12 weeks
  measured using Dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada